CLINICAL TRIAL: NCT04235192
Title: A Multicenter Case-control Study of Risk Factors for Premature Ejaculation in China's Shaanxi Province
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Collaborators: First Affiliated Hospital Xi'an Jiaotong University (Other); Shaanxi Provincial People's Hospital (Other); Xi'an No.3 Hospital (Other Government); Shaanxi Armed Police Corps Hospital (Unknown); Northwest Women's and Children's Hospital, Xi'an, Shaanxi (Other)
Responsible Party: Sponsor
Other Study IDs: 4222018004
Record Dates: First submitted 2020-01-15; First posted 2020-01-21 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Premature Ejaculation
Keywords: risk factor
MeSH Terms: conditions — Premature Ejaculation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Through a multicenter case-control study on the risk factors of premature ejaculation in Shaanxi, to find out the related factors of the occurrence and development of premature ejaculation, to provide reference for personalized treatment, in order to improve the quality of sexual life of patients and partners.

ELIGIBILITY:
Inclusion Criteria:

* 1) case group

  1. 18-64 years old, regular sexual life > 6 months;
  2. Self-report of premature ejaculation;
  3. Able to complete questionnaires and scale scores independently. 2) control group

  <!-- -->

  1. 18-64 years old, regular sexual life > 6 months;
  2. Both partners are satisfied with their sexual life;
  3. Able to complete questionnaires and scale scores independently.

Exclusion Criteria:

* 1) case group

  1. Those who are unable to have sex due to genital malformation;
  2. Patients with serious cardiovascular and cerebrovascular diseases;
  3. Severe mental disorders (history of epilepsy, mania, etc.);
  4. Have a history of brain trauma;
  5. People with a long history of substance abuse. 2) control group

  <!-- -->

  1. Patients with a history of mental illness;
  2. Oral selective serotonin (5-ht) reuptake inhibitors, tricyclic antidepressants, triazolidine antidepressants, tramadol and sedatives

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with premature ejaculation in the outpatient department of the hospital were the case group, while patients without premature ejaculation in the outpatient department were the control group
Sampling Method: Non-Probability Sample
Enrollment: 1340 (Estimated)
Dates: Start 2019-07-31 (Actual); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
IELT | Within 6 months
  Intra-vaginal Ejaculation Latency Time

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital, Fourth Military Medical University, Xi'an, Shaanxi, China